CLINICAL TRIAL: NCT06908200
Title: Effect of Radiofrequency in Women With Chronic Pelvic Pain With an Associated Myofascial Syndrome Versus Myofascial Therapy and no Treatment: a Randomized Clinical Trial
Brief Title: Effect of Radiofrequency in Women With Chronic Pelvic Pain With an Associated Myofascial Syndrome Versus Myofascial Therapy and no Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Carla Box, Principal Investigator, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HCB/2021/0313; HCB/2021/0313 (Other: Ethics Comittee - Hospital Clinic de Barcelona)
Record Dates: First submitted 2025-03-11; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Chronic Pelvic Pain
Keywords: chronic pelvic pain; myofascial syndrome; radiofrequency; manual therapy
MeSH Terms: interventions — Radiofrequency Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ON RF (Active Comparator): Application of the technique in the intervention group (activated resistive capacitive monopolar radiofrequency therapy): the intervention group 1 will receive treatment with activated RF, with the electrode at a medium intensity for 20 minutes per session during a total of 8 sessions, held weekly.
  Interventions: Device: Radiofrequency therapy
- OFF RF (Sham Comparator): Application of the technique in the intervention group (activated resistive capacitive monopolar radiofrequency therapy): the CONTROL group 2 will receive treatment with activated RF, with the electrode for 20 minutes per session during a total of 8 sessions, held weekly.
  Interventions: Device: Radiofrequency therapy
- MYOFASCIAL MANUAL THERAPY (Active Comparator): Application of the technique in the intervention group 2 (MYOFASCIAL MANUAL THERAPY): the intervention group 2 will receive treatment for 20 minutes per session during a total of 8 sessions, held weekly.
  Interventions: Other: myofascial manual therapy
- NO TREATMENT (No Intervention): Patients in waiting list, pending treatment will not receive treatment but symptoms will be monitored after 6 months

INTERVENTIONS:
Device: Radiofrequency therapy — Radiofrequency or myofascial manual therapy sessions including the abdominal region, the vulva and pelvic floor tissue and Thiele massage done daily by the patient at home
  Arms: OFF RF; ON RF
Other: myofascial manual therapy — Myofascial manual therapy sessions including the abdominal region, the vulva and pelvic floor tissue and Thiele massage done daily by the patient at home
  Arms: MYOFASCIAL MANUAL THERAPY

SUMMARY:
A randomised clinical trial is being conducted in the Gynecology Department of the Hospital Clinic de Barcelona in women presenting chronic pelvic pain syndrome due to a myofascial cause which is over a 4 score in the VAS scale and not related to an obstetric injury. This study presents 4 groups; two groups receive 8 radiofrequency sessions, one group receives 8 sessions of myofascial release therapy (MRT) and the last group receives no treatment at all (NT). The two RF groups have been divided into a RF intervention group (RFIG) and a RF control group (RFCG) which receives sham treatment. The RF groups are double-blinded. Other than RF, both groups perform daily Thiele massage at home. The sessions last for 20 minutes and take place once a week during 8 weeks.

The main variable evaluated is the level of pain during the muscular assessment carried out by an expert pelvic floor physical therapist using the Verbal numeric Scale in the first session and at the end of the 8 sessions. Secondary variables are: sexual function (throughout FSFI questionnaire), pain catastrophizing (ECD), quality of life (EQ5D), anxiety and depression (HADS), central sensitization (CSI) as well as other pelvic floor dysfunction symptoms (PFDI).

ELIGIBILITY:
Inclusion criteria included women who were:

* At least 18 years of age
* Presenting with pelvic pain persisting for at least 6 months
* Diagnosed with myofascial syndrome of the pelvic floor muscles (PFM) by a specialist based on physical assessment
* Presenting with pelvic pain intensity greater than 4 on the Visual Analog Scale (VAS) in the last 3 months
* Agreed to sign the informed consent form.

Exclusion criteria included the following:

* Patients who were pregnant
* Postpartum patients who had given birth within the last year
* Patients with a history of vulvovaginal pathology
* Contraindications for the use of radiofrequency: metal implants or active infection
* Patients with a history of pelvic cancer, including those who had undergone chemotherapy, radiotherapy, and/or brachytherapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — WOMEN PRESENTING CHRONIC PELVIC PAIN
Enrollment: 80 (Estimated)
Dates: Start 2022-05-10 (Actual); Primary Completion 2025-06-10 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Pain Level | 8 weeks
  Pain Level using the Verbal Numeric Scale (VNS). The scores go from 0 (lowest) to 10 (highest)

SECONDARY OUTCOMES:
Sexual function | 8 weeks
  Sexual function using the female sexual function index. The score ranges from 2 (severe) to 36 (no sexual disfunction)
Quality of life (QoL) | 8 weeks
  Quality of life using the EuroQuality of life-5Dimensions (EQ5D. Ranges from -0.59 (lowest QoL) and 1 (highest)
Pain catastrophizing | 8 weeks
  Using the pain catastrophizing scale (PCS).Ranges from 0 to 52 where higher scores indicate a greater degree of pain catastrophizing. A total score of >30 represents a clinically significant level of pain catastrophization
Anxiety and depression | 8 weeks
  Anxiety and depression using the Hospital Anxiety and depression Scale (HADS). Generally, scores of 0 to 7 on this questionnaire are considered to be normal, scores of 8 to 10 indicate mild symptoms, 11 to 14 indicate moderate symptoms, and 15 to 21 indicate severe symptoms
Central sensitization | 8 weeks
  Using the central sensitization index (CSI). Ranging from 0-100, >40 is the cutoff for pain sensitization

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No